CLINICAL TRIAL: NCT02699554
Title: Quantifying Patient-Specific Changes in Neuromuscular Control in Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Gillette Children's Specialty Healthcare (Other)
Responsible Party: Principal Investigator, Katherine Steele, Assistant Professor, Mechanical Engineering, University of Washington
Other Study IDs: 44170; 1R01NS091056-01A1 (NIH)
Record Dates: First submitted 2016-01-20; First posted 2016-03-04 (Estimated); Results first posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Orthopaedic surgery
  Interventions: Procedure: Single-event multilevel surgery

INTERVENTIONS:
Procedure: Single-event multilevel surgery

SUMMARY:
Impaired neuromuscular control hinders movement for individuals with cerebral palsy and other neurological disorders. In this research, the investigators are developing new tools to quantify impaired neuromuscular control in cerebral palsy and evaluate changes after one of the most common treatments, orthopaedic surgery. The results from this research will empower clinicians to identify patient-specific factors that contribute to impaired movement and improve treatment and quality of life.

DETAILED DESCRIPTION:
The long-term goals of this research are to quantify patient-specific changes in neuromuscular control in order to optimize treatment planning and improve mobility for individuals with cerebral palsy (CP). As a first step, the aims of this proposal are to evaluate neuromuscular control before and after one of the most common treatments for individuals with CP, orthopaedic surgery. The investigators will evaluate if patient-specific measures of neuromuscular control, based upon the framework of muscle synergies, can predict improvements in walking ability after surgery. Further, investigators will determine whether neuromuscular control changes after surgery and if these changes contribute to improvements in movement. To achieve these goal the investigators will implement and test new tools to quantify neuromuscular control which integrate clinical gait analysis and two computational techniques: synergy analysis and dynamic musculoskeletal simulation. This research will provide the foundation to use measures of altered neuromuscular control to inform treatment planning, develop alternative treatments, and improve mobility in CP and other neurologic disorders.

ELIGIBILITY:
Inclusion Criteria:

* Diplegic cerebral palsy
* Mild or Moderate Impairment, Gross Motor Function Classification System (GMFCS) Levels I-III
* Will receive follow-up care and physical therapy within the Gillette Children's Specialty Healthcare system

Exclusion Criteria:

* Botulinum toxin injections, baclofen, or other similar treatments in the 3 months prior to pre-operative gait analysis

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals with cerebral palsy, diplegia subtype, with mild or moderate impairment, Gross Motor Function Classification System (GMFCS) Levels I-III, between the ages of 6 - 18.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine M Steele, PhD, Principal Investigator — University of Washington
Locations (1):
- Gillette Children's Specialty Healthcare, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 539 children with bilateral cerebral palsy eligible for orthopedic surgery were screened. 122 were invited to participate in the study, 45 did not meet the study criteria, 22 did not respond, and 55 participated in the study.
Groups:
- Orthopaedic Surgery: Single-event multilevel surgery
Period: Overall Study
Arm/Group | Orthopaedic Surgery
Started | 55
Completed | 46
Not Completed | 9
Not completed — Lost to Follow-up | 9

BASELINE CHARACTERISTICS:
Arm/Group | Orthopaedic Surgery
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.5 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 53
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 47
  More than one race | 1
  Unknown or Not Reported | 3
Gait Deviation Index (GDI) [Mean (Standard Deviation); unit: z-score] — normalized z-score such that 100(10) = AVE(SD) of nondisabled peers
  z-score | 68.2 (12.1)
Dynamic Motor Control (DMC) [Mean (Standard Deviation); unit: normalized z-score] | 80.5 (9.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Walk Dynamic Motor Control Index 6-months After Orthopaedic Surgery
Description: The Walk Dynamic Motor Control Index (Walk DMC) is a specific measurement calculated from electromyography during gait using nonnegative matrix factorization. A value of 100 indicates complexity of neuromuscular control similar to typically-developing peers and each 10 point deviation represents one standard deviation from typically-developing peers. Thus, a value of 80 would indicate that an individual's muscle coordination during gait is two standard deviations below the complexity of unimpaired individuals.
Time Frame: 6-months after individual's orthopaedic surgery
Population: 32 of the 55 participants returned for 6-month post-operative gait analysis
Measure: Mean (Standard Deviation); unit: normalized z-score
Arm/Group | Orthopaedic Surgery
Number analyzed (Participants) | 32
normalized z-score | -2.4 (6.0)

2. Primary Outcome: Change in Walk Dynamic Motor Control Index 1-year After Orthopaedic Surgery
Description: as for outcome 1
Time Frame: 1-year after individual's orthopaedic surgery
Population: 46 of the 55 participants returned for 12-month post-operative gait analysis
Measure: Mean (Standard Deviation); unit: normalized z-score
Arm/Group | Orthopaedic Surgery
Number analyzed (Participants) | 46
normalized z-score | -2.7 (6.7)

3. Secondary Outcome: Change in Gait Deviation Index 6-months After Orthopaedic Surgery
Description: The Gait Deviation Index is a specific measurement which uses kinematics measured from instrumented gait analysis to compare an individual's gait pattern to typically-developing controls. A value of 100 indicates kinematics similar to unimpaired individuals while each 10 point deviation represents one standard deviation from unimpaired gait. Thus, a value of 80 would indicate that an individual's gait kinematics are on average two standard deviations from unimpaired gait.
Time Frame: 6-months after individual's orthopaedic surgery
Population: 32 of the 55 participants returned for 6-month post-operative gait analysis
Measure: Mean (Standard Deviation); unit: normalized z-score
Arm/Group | Orthopaedic Surgery
Number analyzed (Participants) | 32
normalized z-score | 2.8 (9.2)

4. Secondary Outcome: Change in Gait Deviation Index 1-year After Orthopaedic Surgery
Description: as for outcome 3
Time Frame: 1-year after individual's orthopaedic surgery
Population: 46 of the 55 participants returned for 12-month post-operative gait analysis
Measure: Mean (Standard Deviation); unit: normalized z-score
Arm/Group | Orthopaedic Surgery
Number analyzed (Participants) | 46
normalized z-score | 2.1 (8.1)

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from baseline to the 12-month follow-up visit.
Arm/Group | Orthopaedic Surgery
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 0/55

LIMITATIONS AND CAVEATS:
This was a prospective observational cohort study, not a randomized controlled trial. 32 of the 55 participants returned for the 6-month post-operative gait analysis and 46 of the 55 participants returned for the 12-month post-operative gait analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT02699554/Prot_SAP_ICF_000.pdf